CLINICAL TRIAL: NCT06546124
Title: Treatment of Upper Trapezius Muscle Myofascial Pain Syndrome: Comparison of Ultrasound- Guided Dry Needling Techniques
Brief Title: Treatment of Upper Trapezius Muscle Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, assistant professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-SK-07
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-09

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep fascia dry needling technique (Active Comparator): Deep fascia dry needling technique
  Interventions: Other: Deep Fascia Dry needling Technique
- İntramuscular trigger point dry needling technique (Active Comparator): İntramuscular trigger point dry needling technique
  Interventions: Other: Intramuscular Trigger Point Dry Needling Technique

INTERVENTIONS:
Other: Deep Fascia Dry needling Technique — "Participants will undergo a single session of dry needling on the painful area of the upper trapezius muscle on the right and/or left side of the neck, either unilaterally or bilaterally. All participants will be positioned upright in a chair with their backs supported, heads in a neutral position, and arms at their sides. A myofascial trigger point on the upper trapezius muscle will be marked. A sterile acupuncture needle, 0.25 mm in diameter and 40 mm in length, will be used. Under ultrasound guidance, the needle will be inserted at three points, including 1 cm lateral and medial to the marked point, penetrating subcutaneously to the deep fascia. After leaving the needle in place for 5 minutes, it will be rotated clockwise and left in place for an additional 5 minutes. The needles will be removed after a total of 10 minutes. Participants will be advised to perform upper trapezius stretching exercises."
  Arms: Deep fascia dry needling technique
Other: Intramuscular Trigger Point Dry Needling Technique — "Participants will undergo a single session of dry needling on the painful area of the upper trapezius muscle on the right and/or left side of the neck, either unilaterally or bilaterally. All participants will be positioned upright in a chair with their backs supported, heads in a neutral position, and arms at their sides. A myofascial trigger point on the upper trapezius muscle will be marked. A sterile acupuncture needle, 0.25 mm in diameter and 40 mm in length, will be used. Under ultrasound guidance, the needle will be inserted at three points, including 1 cm lateral and medial to the marked point, penetrating through the deep fascia into the upper trapezius muscle. After leaving the needle in place for 5 minutes, it will be rotated clockwise and left in place for an additional 5 minutes. The needles will be removed after a total of 10 minutes. Participants will be advised to perform upper trapezius stretching exercises."
  Arms: İntramuscular trigger point dry needling technique

SUMMARY:
The aim of this study is to compare the effects of superficial and deep dry needling techniques, guided by ultrasound, on pain, disability, functional impairment, and quality of life in patients diagnosed with myofascial pain syndrome of the upper trapezius muscle.

DETAILED DESCRIPTION:
Myofascial Pain Syndrome (MAS) is a common condition encountered in the daily practice of musculoskeletal medicine. Dry needling is a commonly used technique by clinicians in the treatment of myofascial trigger points. Dry needling can be classified into two main categories based on the depth of needle insertion: superficial and deep dry needling. Dry needling can be performed using either manual palpation techniques or ultrasonographic imaging. Ultrasound allows for more precise needle placement. It must be recognized that the depth of needling (superficial insertion vs. deep insertion) varies for every structure and that without ultrasound guidance, differentiation between needling into the superficial fascia and beyond the deep fascia maybe difficult. In clinical settings, using ultrasound can help visualize the different layers and guide the needle to the appropriate depth. The aim of this study is to compare the effectiveness of deep fascia and intramuscular trigger point dry needling techniques, guided by ultrasound, on pain, disability, functional impairment, and quality of life in patients diagnosed with myofascial pain syndrome of the upper trapezius muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MPS in the upper trapezius muscle in accordance with criteria defined by Travell and Simons
2. Ages between 20 and 50 years
3. No treatment, including injections, dry needling, and physical methods, applied to the cervical region in the last three months

Exclusion Criteria:

1. Bleeding Tendency
2. History of Neck and Shoulder Trauma
3. Other Conditions Affecting Neck and Shoulder Pain: including malignancy, infection, rheumatic diseases, degenerative joint disease, fibromyalgia, cervical radiculopathy, neuropathy, myelopathy, myopathy, adhesive capsulitis, etc.
4. Cases Where Evaluation Could Not Be Completed for Any Reason
5. Patients Who Refuse to Complete the Evaluations

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-08-11 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The Numerical Pain Rating Scale | Before treatment
  It is used to measure pain. The numerical scale for perceived pain intensity usually includes 11 numbers. The participant selects the number that best reflects their pain. In our study, participants were informed that '0' indicates no pain and '10' represents pain of unbearable intensity.
The Numerical Pain Rating Scale | 1 week after treatment
  It is used to measure pain. The numerical scale for perceived pain intensity usually includes 11 numbers. The participant selects the number that best reflects their pain. In our study, participants were informed that '0' indicates no pain and '10' represents pain of unbearable intensity.
Pressure Pain Threshold | Before treatment
  A pressure algometer (dolorimeter) is a device used for assessing pain sensitivity and measuring pressure perception. It has been proven useful in evaluating trigger points, arthritis activation, and visceral pain-pressure sensitivity. The pressure algometer consists of a metal piston with a rubber disc at the end, which has a 1 cm² surface, and is connected to a gauge that measures pressure in kilograms of force (kgf). In our study, a manual algometer (Baseline® Dolorimeter, Fabrication Enterprises, Inc, NY, USA) was used. The algometric measurement will be performed three times on the most painful point as reported by the patient and detected by palpation. The average of these three measurements will be included in the evaluation.
Pressure Pain Threshold | 1 week after treatment
  A pressure algometer (dolorimeter) is a device used for assessing pain sensitivity and measuring pressure perception. It has been proven useful in evaluating trigger points, arthritis activation, and visceral pain-pressure sensitivity. The pressure algometer consists of a metal piston with a rubber disc at the end, which has a 1 cm² surface, and is connected to a gauge that measures pressure in kilograms of force (kgf). In our study, a manual algometer (Baseline® Dolorimeter, Fabrication Enterprises, Inc, NY, USA) was used. The algometric measurement will be performed three times on the most painful point as reported by the patient and detected by palpation. The average of these three measurements will be included in the evaluation.
Neck disability index | Before treatment
  The Neck Disability Index (NDI) Turkish version was used for assessing patients' disability. This index is a scale consisting of 10 questions used to evaluate how and to what extent neck pain affects the patient's daily living activities. The scale includes parameters such as pain intensity, self-care, lifting, reading, headache, concentration, driving, sleep, and social activities. Patients were asked to mark the option that best applies to them from the 6 choices provided for each parameter. Each item is scored from 0 (no disability) to 5 (complete disability). The total score ranges from 0 (no disability) to 50 (total disability). After obtaining the total score, the value calculated according to the formula is expressed as a percentage of impairment. As the score increases, disability increases; as the score decreases, disability decreases.
Neck disability index | 1 week after treatment
  The Neck Disability Index (NDI) Turkish version was used for assessing patients' disability. This index is a scale consisting of 10 questions used to evaluate how and to what extent neck pain affects the patient's daily living activities. The scale includes parameters such as pain intensity, self-care, lifting, reading, headache, concentration, driving, sleep, and social activities. Patients were asked to mark the option that best applies to them from the 6 choices provided for each parameter. Each item is scored from 0 (no disability) to 5 (complete disability). The total score ranges from 0 (no disability) to 50 (total disability). After obtaining the total score, the value calculated according to the formula is expressed as a percentage of impairment. As the score increases, disability increases; as the score decreases, disability decreases.
Neck bournemouth questionnaire | Before treatment
  Adapted from the Bournemouth Low Back Pain Questionnaire developed by Bolton and Humphreys in 2002, this questionnaire includes variables that must be assessed in individuals with neck pain. The content of the questionnaire covers pain intensity, the impact of pain on daily living activities and social life, anxiety and depression levels, kinesiophobia, and pain coping strategies. Each of the 7 questions is scored from 0 to 10. The highest possible score is 70, with a higher score indicating a higher level of disability.
Neck bournemouth questionnaire | 1 week after treatment
  Adapted from the Bournemouth Low Back Pain Questionnaire developed by Bolton and Humphreys in 2002, this questionnaire includes variables that must be assessed in individuals with neck pain. The content of the questionnaire covers pain intensity, the impact of pain on daily living activities and social life, anxiety and depression levels, kinesiophobia, and pain coping strategies. Each of the 7 questions is scored from 0 to 10. The highest possible score is 70, with a higher score indicating a higher level of disability.
Joint range of Motion Measurement | Before treatment
  Joint range of motion is measured using a goniometric protractor with the Neutral-0 Method. While the person sits upright in a chair, the goniometer is used to measure the range of motion of the neck in the directions of flexion, extension, lateral flexion, and rotation.
Joint range of Motion Measurement | 1 week after treatment
  Joint range of motion is measured using a goniometric protractor with the Neutral-0 Method. While the person sits upright in a chair, the goniometer is used to measure the range of motion of the neck in the directions of flexion, extension, lateral flexion, and rotation.

SECONDARY OUTCOMES:
Advers event | 1 week after treatment
  Follow-up will include assessment of pain-burning sensation, nausea, dizziness, and pain experienced during the procedure.
Cutaneous and subcutaneous thickness | Before treatment
  Cutaneous and subcutaneous tissue thickness will be measured with ultrasound at the site of the trigger point in the upper trapezius muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No